CLINICAL TRIAL: NCT05526547
Title: Implant-supported Zirconia Fixed Partial Dentures Cantilevered in the Lateral-posterior Area
Brief Title: Implant-supported Zirconia Partial Dentures With Cantilever
Status: Completed | Type: Observational
Sponsor: D'Albis Dental (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, D'Albis Dental
Other Study IDs: cantilever
Record Dates: First submitted 2022-08-26; First posted 2022-09-02 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Fifteen partially edentulous patients received 34 implants and were provided 16 zirconia fixed partial prostheses (FPPs) with one cantilever extension replacing mandibular or maxillary missing posterior and lateral teeth. Patients were re-examined up to 4 years.

DETAILED DESCRIPTION:
The investigators consecutively enrolled 15 patients who required dental implant rehabilitation with fixed dental prosthesis. All patients were attended at a private out-patient clinic from 2018 to 2021.The study was conducted in Italy and all procedures respect European laws and regulations.A diagnostic wax-up of the missing teeth was performed on digital casts for each case. Each case was designed using software planning the implant position in the distal part of the edentulous ridge where the bone conditions were more favorable.The surgical procedures were performed according to the protocols given by manufacturers.The implant site was prepared after raising a full-thickness flap. The implant was placed as designed in the digital planning with the support of a surgical guide.The patients were recalled 3-6 months after surgery for a pre-prosthetic evaluation. A healing abutment was placed, and implant stability was proven.Three weeks after second-stage surgery, the definitive digital impression was taken using an intraoral scanner. The prosthetic procedures were performed according to manufacturers' implant system recommendations. All prostheses were designed using CAD software with a connector cross-sectional area of at least 12 mm2. Monolithic zirconia fixed partial dentures were fabricated using a CAD-CAM unit from pre-sintered, pre-shade zirconia blanks . The fixed dentures were characterized with ceramic-based colors. The screw-retained zirconia prosthesis were subsequently inserted, and a check of the occlusion was performed.The patients get a baseline examination after 1-3 weeks of final prosthesis insertion. Aesthetics, proximal contacts, and occlusion were modified when needed following a careful examination. Patients were recalled at least once a year to assess the restorations functionally and aesthetically, peri-implant tissues, and implant health status. An individual maintenance program with regular dental hygiene sessions was performed during the entire study period for every patient, and an x-ray was taken at the 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Good health according to the System of the American Society of Anesthesiology
* Aged older than 18 years
* No general medical contraindication for implant therapy
* Two or more missing teeth from the canine to the second molar
* Good periodontal health or treated periodontitis

Exclusion Criteria:

* Smoking more than 15 cigarettes a day
* Untreated periodontitis
* Pregnancy
* Acute infections
* Keratinized mucosal tissue less than 2 mm.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who required dental implant rehabilitation with fixed dental prostheses.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prosthesis | 4 years
  Evaluation of prosthetic clinical complication of the Fixed Partial Dentures: zirconia chipping (yes or not), zirconia Fracture (yes or not) , loosening of abutment screw (yes or not).

SECONDARY OUTCOMES:
Implant | 4 years
  Evaluation of biological complication implants related. Clinical outcome: mucositis(yes or not: blending on probing) , periimplantitis (yes or not: supuration and 3mm at least of marginal bone loosening), implants fractures (yes or not).

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe D'Albis, Mola di Bari, Bari, Italy